CLINICAL TRIAL: NCT01322932
Title: HIV-positive Patients Under Tenofovir, Emtricitabine and Efavirenz Therapy Switching From a Two-pill Regimen to a Single Pill Regimen: Patients'Opinion Survey
Brief Title: Tenofovir, Emtricitabine and Efavirenz Late Switch to a Single Pill: Patients' Opinion Survey
Status: Completed | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Swiss HIV Cohort Study (Network); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Marie Schneider, Pharmacist, PhD, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Other Study IDs: 151/10
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infection
Keywords: Medication Adherence; HIV Infection; efavirenz, emtricitabine, tenofovir disoproxil fumarate drug combination [Substance Name]; efavirenz; emtricitabine; Patient Satisfaction; tenofovir disoproxil fumarate
MeSH Terms: conditions — HIV Infections; Medication Adherence; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess adherence, tolerability and satisfaction of each eligible HIV subjects switching from a two- or three-pill tenofovir-emtricitabine-efavirenz (TDF-FTC-EFV) to a one-pill TDF-FTC-EFV treatment.

DETAILED DESCRIPTION:
Each eligible patient will be screened from de SHCS database. Each refusal and drop-out will be documented. A pre-visit (V-1) will be scheduled for informed consent, V0 for inclusion (V-1 and V0 may occur on the same day), V1 one month post-inclusion and V2 4 to 7 months post-inclusion. V0, V1 and V2 will be planned during regular medical visits.

Eligible patients either get their cART in their usual pharmacy according to standard of care, or take part in a routine adherence-enhancing program(adherence subgroup)run by the pharmacists of the outpatient medical clinic.

In the adherence subgroup, adherence is assessed electronically by MEMS (Medication event monitoring system) monitors on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* patients under TDF-FTC-EFV
* followed up at the Service of Infectious Disease of the University Hospital of Lausanne
* enrolled in the SHCS

Exclusion Criteria:

* patients receiving TDF-FTC-EFV in combination with other ARTs
* patients under TDF-FTC-EFV for less than 3 months
* patients not fluent in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under TDF-FTC-EFV followed up at the Service of Infectious Disease of the University Hospital of Lausanne and enrolled in the Swiss HIV Cohort Study (SHCS) Adherence subgroup: patients enrolled in the HIV adherence program at the pharmacy of the Department of Ambulatory Care & Community Medicine in Lausanne.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Patient adherence | V0, V1, V2
  by questionnaire in both subgroups and by MEMS data in the adherence subgroup
Adverse events and symptoms | V0, V1, V2
  by questionnaires
Treatment management | V0, V1, V2
  Treatment management according to meals, timing, disruptive daily schedule By questionnaire
Patient satisfaction of the switch | V1, V2
  By questionnaire

SECONDARY OUTCOMES:
Impact of switch on clinical outcomes | V0, V1, V2
  Clincal outcomes = viral load, CD4 count, resistance, EFV blood level. By medical file
Patients' acceptance of switch | V-1

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Cavassini, M.D, Study Chair — Centre Hospitalier Universitaire Vaudois; Marie-Paule Schneider, PhD, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Olivier Bugnon, Professor, Study Chair — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Aurélie Gertsch, PhD Student, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Locations (1):
- Centre Hospitalier Universitaire Vaudois et Policlinique Medicale Universitaire, Lausanne, Canton of Vaud, Switzerland